CLINICAL TRIAL: NCT04549688
Title: Active Surveillance Plus (AS+): Local Tumor Control With High-intensity Focused Ultrasound (HIFU) in Patients With Localized Prostate Cancer
Brief Title: Active Surveillance Plus (AS+): High-intensity Focused Ultrasound (HIFU) in Patients With Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Sven Löffeler, Principal Investigator, The Hospital of Vestfold
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS-plus-SiV-01
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; HIFU; focal treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: prospective, single-arm, case-control cohort study with consecutive patients with intermediate-risk, MRI-visible prostate cancer treated focally with HIFU. Study patients will be compared to historical controls (patients observed with AS at SiV 2009-2017).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focal therapy (Experimental)
  Interventions: Procedure: high-intensity focused ultrasound, HIFU

INTERVENTIONS:
Procedure: high-intensity focused ultrasound, HIFU — see above

SUMMARY:
PSA (Prostate-specific antigen) testing has significantly increased the number of men diagnosed with prostate cancer (PCa) and especially patients with low and intermediate risk disease. The effect of radical treatment (treatment of the entire prostate gland) in these risk groups is disputable while the risk of adverse effects, with erectile dysfunction and urinary incontinence, is not. Active surveillance (AS) has been developed as an alternative to radical treatment with the aim of avoiding or delaying radical treatment by closely monitoring for signs of tumor progression. Active surveillance is regarded as the treatment of choice for low-risk prostate cancer. Focal therapy may have a crucial role in improving active surveillance protocols for patients with intermediate localized prostate cancer. Focal eradication of the index-tumor may delay or avoid indefinitely radical treatment for this patient group while significantly reducing treatment-related side effects. Improved MRI-diagnostics and MRI/ ultrasound fusion technology have optimized tumor mapping and classification and this in turn has made partial treatment of the prostate a feasible treatment option.

This study is a prospective cohort study. Patients with intermediate (high-risk) localized PCa and a visible index tumor will be treated with high-intensity focused ultrasound (HIFU).

The aim of the study is to show that there is a significant effect of focal treatment on surveillance biopsies and a reduced conversion to radical treatment, without compromising survival outcomes compared to historical controls (retrospective cohort). A cohort from the more than 450 patients included in the local AS-protocol with MRI at Vestfold hospital trust since 2009 will serve as controls.

DETAILED DESCRIPTION:
1 Needs description It is unclear if eradication with focal treatment of the index-tumor of patients with intermediate-risk prostate cancer followed by active surveillance can reduce the need for radical, whole-gland treatment of the prostate and thereby treatment side effects. It is important for urologists and patients to know if focal treatment of prostate cancer is both a safe and effective treatment option. If proven so, focal treatment of prostate cancer can be offered as a viable, intermediate treatment option for a large group of patients who currently only have the choice between either surveillance or radical treatment.

Thus, there is an unmet need to document the outcome of focal treatment in selected patients with prostate cancer, both in terms of efficacy and safety

2. Hypotheses, aims and objectives

2.1 Hypothesis: Focal treatment of biopsy-verified, localized, MRI-visible, intermediate-risk (and high-risk fo elderly patients) prostate cancer is a safe and effective treatment option. Side effects following focal treatment are transient and mild compared to established and well-documented radical treatment options.

2.2 Aims of the study: To investigate if focal treatment of localized prostate cancer followed by MRI-supplemented active surveillance conveys sufficient tumor control to enable patients to continue indefinitely in this follow-up protocol without the need to convert to radical treatment, with none or mild side effects and without compromising oncological outcomes.

2.3 Objectives:

Primary objectives:

* Eradication of the signal tumor (<20% positive biopsies in the treated area after one year)
* Low conversion rates to radical treatment (<20%)
* Good long-term oncological results (<5% metastasis and <1% prostate cancer deaths at 10 years)
* Good functional results (<10% of patients with long-term side effects on erectile function and continence)

Secondary objectives:

* Evaluation of the ability of MRI to predict biopsy results during follow-up.
* Health-related quality of life

  3. Methodology

This study is a prospective, single-arm, case-control cohort study with consecutive patients with intermediate-risk, MRI-visible prostate cancer treated focally with HIFU. Participants will be compared to historical controls (patients observed with AS at SiV 2009-2017). The study design follows the international multidisciplinary consensus on trial design for focal therapy in PCa (28, 29). Patients will primarily be recruited from Vestfold-Telemark County but recruitment from other institutions in Norway is encouraged. More formal referral arrangements will be sought with Aleris (Oslo), Telemark Hospital Trust and Vestre Viken Hospital Trust.

3.1 Project arrangements, method selection and analyses From a scientific and methodological point of view a randomized, parallel-group study would have been preferable with patients receiving either AS+ (HIFU) or simple AS follow-up. However, experience from several investigative centers have shown that randomization is difficult to carry out in practice. This is because patients are aware of the HIFU possibility, and, if randomized to standard treatment, often refuse participation and demand HIFU treatment. This problem would likely be exacerbated in this study, where the control group would be offered only follow-up while study arm patients receive tumor-directed treatment with presumed few side-effects. Furthermore, the investigators have learned from own historic controls that AS is "good medicine" for merely half of the patients with intermediate-risk prostate cancer after 5 years. Since it is difficult, based on today's diagnostic tools, to identify patients that will not progress significantly over time, some form of tumor-directed treatment for all patients is sensible. Finally, patients in the historical control group were diagnosed and risk-classified by the same parameters and diagnostic tools that are currently in use. Follow-up of these patients was also very similar to the one outlined for the study patients. The investigators are not aware of any significant change in clinical practice that would suggest that the historical controls at the study institution are not representative of current patients with intermediate risk profile.

Patients who are interested in focal treatment of prostate cancer are aware of the radical treatment alternatives but are skeptical of the side effects. These patients want to know their risk of progression (metastasis and death), the risk of having to undergo radical treatment at a later stage and the short-term and long-term side effects if they choose focal treatment. We believe that this study will provide these answers for a representative Norwegian patient population.

Based on these considerations, the investigators believe that the best and most ethical design is the one proposed here, where all eligible patients receive the same treatment and are then compared to a historical control group.

Study population and Power-estimate Approximately half of active surveillance patients (50%) experience progression of their disease during 5-10 years follow-up (9). This correlates with the outcome of historical AS patients at the study institution.

The investigators estimate that only 20% of the newly diagnosed AS patients receiving HIFU will experience a progression of their disease after 10 years.

In order to detect such a reduction in progression rate, the trial will need to include 194 patients. With 20% expected dropouts, the number of patients needed to include in the HIFU cohort will be 245.

The sample size calculations are based on the ClinCalc program (http://clincalc.com/stats/samplesize.aspx).

ELIGIBILITY:
Inclusion Criteria:

* Age 55-80 years
* Life expectancy >10 years
* Gleason-score:

  * patients <75 years: Gleason score < 8
  * patients 75-80 years: Gleason <9
* TNM-stage: clinical/ radiological stage <T2c (localized), rN0 and rM0
* PSA < 15
* PSA > 15 should be counseled with caution (does not apply to patients >75 years)
* Risk group: d'Amico intermediary risk group, open for high risk patients age >75 years

Exclusion Criteria:

* Previous treatment
* Previous treatment of the primary cancer within the prostate
* Previous hormone treatment for prostate cancer within 6 months before trial
* Previous radiation to pelvis
* Acute urinary tract infection
* For patients <75 years: >5% chance of lymph node metastases calculated by the updated prostate cancer staging nomogram (Partin tables) (30)
* Radiological imaging:
* PI-RADS score <3, clinical significant cancer is equivocal
* Extracapsular extension or seminal vesicle invasion
* Lymph node or bone metastasis
* > 2 MRI detected tumors validated by systematic or MRI-guided biopsies
* Contraindications for MRI

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male prostate cancer patients
Enrollment: 250 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients without clinically significant prostate cancer | 1-10 years
  Absence of clinically significant prostate cancer (Gleason grade ≥7A) on post-treatment systematic and targeted biopsies
Measurement of functional results | 1-10 years
  erectile function, continence, and other therapy-related complications. Questionnaire-based.
Number of patients who need repeated focal treatment | 1-10 years
  recurrence and recurrent treatment
Number of patients eligible for continuous AS+ | 1-10 years
Disease-free survival | 1-10 years
  based on repeated MRI and repeat biopsies performed on clinical/ radiological suspicion
Treatment-free survival | 1-10 years
Overall survival | 1-10 years
Metastasis-free survival | 1-10 years
Number of patients who need radical (surgery or radiation), or palliative treatment (hormone therapy) | 1-10 years

SECONDARY OUTCOMES:
Number of patients where MRI predicted tumor recurrence/ tumor absence | 1-10 years
  MRI findings verified by biopsies
Patient Reported Outcomes Measures | 1-10 years
  Survey-based using standard questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Sven Löffeler, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Vestfold Hospital Trust (Hospital of Vestfold), Tønsberg, Vestfold, Norway

IPD SHARING:
Plan to Share IPD: No